CLINICAL TRIAL: NCT01715961
Title: Multicentric Prospective Study to Assess the Clinical and Prognostic Value of Sarcopenia in Patients Older Than 70 Years With Diffuse Large B-cell Lymphoma
Brief Title: Clinical and Prognostic Value of Sarcopenia in Patients Older Than 70 Years With Diffuse Large B-cell Lymphoma
Acronym: SARCOPENIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHB 11-02
Record Dates: First submitted 2012-04-11; First posted 2012-10-29 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-07

CONDITIONS: Diffuse Large B Cell Lymphoma; Grade IIIB Follicular Lymphoma
Keywords: 70 years old; DLBCL; Rituximab-CHOP; Sarcopenia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anthropometric measurement (Other): The muscle area assessed by CT scan imaging at a lumbar vertebral landmark (L3) at the time of diagnosis, at the end of treatment, at 12 and 18 months
  * anthropometric measures (weight, height, BMI, brachial and calf circumference) and MNA (mini nutritional assessment)
  * albuminemia, transthyretin, orosomucoid, CRP
  * functional test to attest the muscular strength: hand grip test, unipodal test, up and go test
  * hematological and non-hematological chemotherapy toxicities of cycle 1 and cycle 2
  * OS and PFS at 18 and 24 months
  * GCB and ABC phenotypes determined by immunohistochemistry and transcriptome analysis
  Interventions: Procedure: anthropometric measurement

INTERVENTIONS:
Procedure: anthropometric measurement — To attest the muscular strength: hand grip test, balance test, up and go test
  Other Names: Hand Grip strength test; Timed get up and go test

SUMMARY:
This clinical trial is a multicentric prospective study to assess the clinical and prognostic value of sarcopenia in patients older than 70 years with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Sarcopenia status is assessed by CT scan imaging on the overall survival at 18 months in patients older than 70 years with diffuse large B-cell lymphoma treated by R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 70 years
* DLBCL, grade IIIB follicular lymphoma or histologically proven transformed low grade lymphoma
* Whatever the IPI score and the performance status
* Treated by Rituximab-CHOP or Rituximab-mini-CHOP
* CT scan imaging performed one month or less before inclusion
* Signed informed consent

Exclusion Criteria:

* No initial CT scan imaging performed more than one month before inclusion
* Positivity for HCV, HBV and HIV
* Anthracycline contra-indication

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
progression free survival | at 18 months

SECONDARY OUTCOMES:
progression free survival | at 24 months
rate of over grade 2 toxicities | at the first and second courses of chemotherapy (day 21 and day 42)
determination of both molecular subtypes GCB and ABC | at 24 months
  according DASL technology (c-DNA mediated annealing selection extension and ligation)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice JARDIN, MD;PhD, Study Director — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No